CLINICAL TRIAL: NCT01856673
Title: Evaluation of Two Mental Health Interventions Based on the Community for Violence-Displaced Afro-Descendants in Colombia.
Brief Title: Evaluation of Two Community-based Mental Health Interventions for Violence-Displaced Afro-Descendants in Colombia.
Acronym: ACOPLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Valle, Colombia (Other)
Collaborators: Heartland Alliance (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Johns Hopkins Bloomberg School of Public Health (Other); Afrocolombian Displaced Association - AFRODES (Unknown)
Responsible Party: Principal Investigator, Maria Isabel Gutiérrez Martínez, Professor, Universidad del Valle, Colombia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HA-UV-JHU-2013-001; U1111-1138-4894 (Registry Identifier: Universal Trial Number (UTN))
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Post-Traumatic Stress Disorder; Depression; Anxiety; Violence
Keywords: Mental Health; Displacement; Torture; Violence; Post-Traumatic Stress Disorder; Depression; Anxiety; Community-based intervention; Prevention trial; Disabled Persons
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ARM 1: Component-Based Intervention (Experimental): Common Elements Treatment Approach (CETA) only
  Interventions: Behavioral: Common Elements Treatment Approach
- ARM 2: Community Group Therapy (Experimental): Narrative Community Group Therapy (NCGT) only
  Interventions: Behavioral: Narrative Community Group Therapy
- ARM 3: Standby group (Other): Standby group without intervention, but under monthly monitoring.
  Interventions: Other: Standby group

INTERVENTIONS:
Behavioral: Common Elements Treatment Approach — It was developed for treating symptoms related to violent trauma, i.e. symptoms of depression, anxiety and distress, among a population victimized by violence and torture in Colombia. The most relevant components for treatment of these 3 problematic issues were identified from literature review and a panel of experts. Descriptions and schemes have been developed in order to guarantee facility of use by community counselors who have little background in mental health skills. These counselors, who will be called Lay Psychosocial Community Workers (LPCW), will receive training in this technique before beginning of interventions. Application of this technique will be supervised constantly by mental health professionals (psychologist or social worker) from the project team.
  Other Names: CETA
  Arms: ARM 1: Component-Based Intervention
Behavioral: Narrative Community Group Therapy — It consists on teaching skills to people in the community to provide mental health therapy. Therapy will be performed by LPCW under constant supervision of mental health professionals (psychologists or social workers). Sessions will begin with a series of introductory activities that motivates participants to propose different problems that they would like to solve in the group. A participant proposed a problem and he/she will be asked to talk about it. LPCW and/or psychologist will support individuals if anyone needs help to solve a psychological crisis. At the end of this narration, participants will be asked about who has had a similar situation, and how they solved it. In this way, proposed solutions will be collected by the LPCW. Finally, session closes with a motivating activity.
  Other Names: NCGT
  Arms: ARM 2: Community Group Therapy
Other: Standby group — Standby group: they will be assessed at baseline with the initial survey and they will wait between 10 and 12 weeks; an exit assessment will be performed with the study instrument. After the exit survey, control group participants will have an appointment with a professional psychologist to determine whether they require a mental health treatment. Those with such necessity will receive treatment in the ACOPLE center by professional psychologists or they will be referred to other health care level according to the type of psychopathology (e.g., psychosis) or its severity. Also, participants in the control group will be monitoring monthly by phone calls and if they have any psychological problem, they will be assessed in the ACOPLE center.
  Arms: ARM 3: Standby group

SUMMARY:
This study is a community prevention randomized trial with three parallel groups: two intervention groups and one control group in Buenaventura and Quibdó.

The aim of the trial is to evaluate the impact of two community interventions on mental health; the intervention groups are designed to decrease depression, anxiety, post-traumatic stress disorders symptoms as well as the level of dysfunctionality in Afro-Colombian victims of violence.

Adult people (equal or more than 18 years old) belonging to Afro-Colombian communities in both cities will participate in the enter survey. The subjects will be selected based on the severity of symptoms, traumatic experiences and a level of dysfunction identified using the instruments of this research (i.e. those obtaining an score equal or higher than 49 in symptoms (25% of the total of symptoms)).

The fieldwork and the interventions will be conducted by people belonging to the community; they are called Lay Psychosocial Community Workers (LPCW). After six (6) weeks of formal training, they will be able to perform two kinds of interventions, Common Elements Treatment Approach (CETA) based on a cognitive behavioral intervention and Narrative Community Group Therapy (NCGT), for the people affected by violence and displacement that were pre-selected according to the baseline instrument.

The LPCW will be under the constant supervision by psychologists of the project, and under weekly supervision by a group of experts from Johns Hopkins University, the Heartland Alliance and The Institute for Research and Development in Violence Prevention and Promotion of Peaceful Coexistence Social (CISALVA) by means of phone calls or monthly visits to the cities. Selected subjects will be randomly allocated to any study branch: CETA, NCGT or the waiting control group.

The study subjects will follow their allocated treatment, or waiting in the control group, for 8 to 12 weeks; then they will be re-assessed using the project instrument two weeks after the last session of therapy.

The study outcome is the differences in instrument scores between the follow-up and the baseline among the interventions (CETA or NCGT) and control group.

Control subjects will be assessed by the project psychologist after the follow-up, and they will receive treatment when necessary.

DETAILED DESCRIPTION:
Colombian armed conflict predominantly affects rural communities; armed conflict has caused thousands of deaths and the displacement of a vast amount of people from rural areas. A considerable amount of the displacement comes from the two most important cities in Pacific coast region: Buenaventura in Valle del Cauca province and Quibdó in Chocó province.

This project will assess treatments, Common Elements Treatment Approach (CETA) and Narrative Community Group Therapy (NCGT), to reduce mental symptoms triggered by violence and will develop mechanisms for a sustainable supply of mental health services in the region.

Adult Afro-Colombian persons who have responded to the study survey but present symptoms of severe mental illness like schizophrenic, psychotic, suicidal attempters, those who can potentially harm others, or who require specialized treatment will not be included in the study.

They will be referred to a project psychologist who will determine whether they require psychiatric treatment, in which case, they will be referred to health institutions through social workers who will ensure treatment is given. Finally, anyone who is related to the LPCW will be excluded.

For the CETA arm, new clients will be enrolled as long as a treatment position becomes available (i.e., as long as previous clients have completed the treatment) to keep the providers (LPCW) running at full capacity. These new clients will be chosen from those randomly allocated to receive the CETA treatment; within fifteen (15) days of the completion of treatment the participants will be reassessed.

Similarly, the NCGT arm will form new groups as long as place becomes available (i.e, as long as previous group has finished treatment) to keep providers running at full capacity. Group members will be chosen from randomly allocated participant to receive NCGT, selecting enough people each time to fill up a group before the treatment begins. All group members will be reassessed within fifteen (15) days of completing the NCGT.

The participants allocated in the control group will undergo a waiting period similar to the period between the initial and final assessments of those receiving CETA and NCGT. This period is estimated to be 3 months, but it could be longer if there are treatment delays. At the end of this time, the participants will be reassessed.

after the control group is reassessed they will be evaluated and receive professional attention by psychologists to decide what is the best intervention that we can offer to the clients in both cities.

Missing values will be handle using multiple imputation methods and data will be analyzed with an intention to treat basis. Sensitivity analysis will be carried out using non-imputed database and including co-variables in the models the inverse probability weight to lost of follow-up.

The anticipated results is a reduction in anxiety, depression and post-traumatic stress disorder symptoms of 20 points among subjects in intervention groups (CETA or NCGT ) compared with those in the control group.

An adherence of 70% is expected to generate strategies for the promotion and prevention in mental health for Afro-Colombian victims of violence and displacement.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older) Afro-Colombian victims of violence and torture who have expressed sadness, suffering psychological trauma caused by violence and when the situation was known by the leaders of Afro-Colombian Displaced Association (AFRODES) or the community leaders contacted by the research team.
* Persons with a total symptomatic value greater than or equal to 49 points in the study instrument, with the presence of trauma from violence, and a loss of functionality score greater than zero.
* Individuals who signed the informed consent.

Exclusion Criteria:

* People of ethnicities other than Afro-Colombian.
* Children under 18 years old.
* Persons who present symptoms of severe mental illness such as schizophrenia, psychotic episodes, suicidal attempters, and those who potentially could harm others.
* Anyone who is related with the counselors (LPCW).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: María Isabel Gutiérrez Martínez, MD, MSc, PhD, Study Director — CISALVA Institute of Universidad del Valle, Colombia; Andrés Fandiño Losada, MD, MSc, PhD, Principal Investigator — CISALVA Institute of Universidad del Valle, Colombia; Francisco Javier Bonilla Escobar, MD, MSc, Principal Investigator — CISALVA Institute of Universidad del Valle, Colombia; Diana Milena Martínez Buitrago, MD, MSc, Principal Investigator — CISALVA Institute of Universidad del Valle, Colombia; Julián Santaella, VMD, MSc, Principal Investigator — CISALVA Institute of Universidad del Valle, Colombia
Locations (2):
- Colombia (2):
  - Centro ACOPLE de Quibdó, Quibdó, Departamento del Chocó
  - Centro ACOPLE de Buenaventura, Buenaventura, Valle del Cauca Department

REFERENCES:
- [Background] Sjolund BH, Kastrup M, Montgomery E, Persson AL. Rehabilitating torture survivors. J Rehabil Med. 2009 Sep;41(9):689-96. doi: 10.2340/16501977-0426. PMID 19774300
- [Background] Bisson J, Andrew M. Psychological treatment of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003388. doi: 10.1002/14651858.CD003388.pub3. PMID 17636720
- [Background] Kinzie JD. Psychotherapy for massively traumatized refugees: the therapist variable. Am J Psychother. 2001;55(4):475-90. doi: 10.1176/appi.psychotherapy.2001.55.4.475. PMID 11824215
- [Result] Murray LK, Tol W, Jordans M, Zangana GS, Amin AM, Bolton P, Bass J, Bonilla-Escobar FJ, Thornicroft G. Dissemination and implementation of evidence based, mental health interventions in post conflict, low resource settings. Intervention (Amstelveen). 2014 Dec;12(Suppl 1):94-112. doi: 10.1097/WTF.0000000000000070. PMID 28316559
- [Result] Osorio-Cuellar GV, Pacichana-Quinayaz SG, Bonilla-Escobar FJ, Fandino-Losada A, Gutierrez-Martinez MI. Perceptions about implementation of a Narrative Community-based Group Therapy for Afro-Colombians victims of Violence. Cien Saude Colet. 2017 Sep;22(9):3045-3052. doi: 10.1590/1413-81232017229.00402016. PMID 28954155
- [Result] Pacichana-Quinayaz SG, Osorio-Cuellar GV, Bonilla-Escobar FJ, Fandino-Losada A, Gutierrez-Martinez MI. Common Elements Treatment Approach based on a Cognitive Behavioral Intervention: implementation in the Colombian Pacific. Cien Saude Colet. 2016 Jun;21(6):1947-56. doi: 10.1590/1413-81232015216.07062015. PMID 27276543
- [Result] Bonilla-Escobar FJ, Osorio-Cuellar GV, Pacichana-Quinayaz SG, Sanchez-Renteria G, Fandino-Losada A, Gutierrez MI. Do not forget culture when implementing mental health interventions for violence survivors. Cien Saude Colet. 2017 Sep;22(9):3053-3059. doi: 10.1590/1413-81232017229.12982016. PMID 28954156
- [Result] Bonilla-Escobar FJ, Fandino-Losada A, Martinez-Buitrago DM, Santaella-Tenorio J, Tobon-Garcia D, Munoz-Morales EJ, Escobar-Roldan ID, Babcock L, Duarte-Davidson E, Bass JK, Murray LK, Dorsey S, Gutierrez-Martinez MI, Bolton P. A randomized controlled trial of a transdiagnostic cognitive-behavioral intervention for Afro-descendants' survivors of systemic violence in Colombia. PLoS One. 2018 Dec 10;13(12):e0208483. doi: 10.1371/journal.pone.0208483. eCollection 2018. PMID 30532155
- [Result] Bonilla-Escobar FJ, Lim HM. A Call for Action for Mental Health: Medical Students and Physicians' roles. International Journal of Medical Students. 2015;3(3):121-122. https://doi.org/10.5195/ijms.2015.131
- [Result] Pacichana-Quinayaz SG, Osorio-Cuellar GV, Gonzalez S, Bonilla-Escobar FJ, Gutierrez-Martinez MI. Relevance of Qualitative Research Approach in Evaluating Mental Health Interventions among Victims of Violence. International Journal of Medica Students. 2015;3(3):170-171. https://doi.org/10.5195/ijms.2015.194
- [Result] Santaella-Tenorio J, Bonilla-Escobar FJ, Nieto-Gil L, Fandino-Losada A, Gutierrez-Martinez MI, Bass J, Bolton P. Mental Health and Psychosocial Problems and Needs of Violence Survivors in the Colombian Pacific Coast: A Qualitative Study in Buenaventura and Quibdo. Prehosp Disaster Med. 2018 Dec;33(6):567-574. doi: 10.1017/S1049023X18000523. Epub 2018 Jul 26. PMID 30047356
- [Derived] Bonilla-Escobar FJ, Fandino-Losada A, Martinez-Buitrago DM, Santaella-Tenorio J, Escobar-Roldan I, Tobon-Garcia D, Munoz-Morales EJ, Babcock L, Duarte-Davidson E, Murray LK, Gutierrez-Martinez MI. Mental health Narrative Community-Based Group Therapy in violence-displaced Afro-Colombians: a randomized controlled trial. Med Confl Surviv. 2023 Mar;39(1):28-47. doi: 10.1080/13623699.2023.2177951. Epub 2023 Feb 23. PMID 36815261
- [Derived] Bonilla-Escobar FJ, Osorio-Cuellar GV, Pacichana-Quinayaz SG, Rangel-Gomez AN, Gomes-Pereira LD, Fandino-Losada A, Gutierrez-Martinez MI. Impacts of violence on the mental health of Afro-descendant survivors in Colombia. Med Confl Surviv. 2021 Jun;37(2):124-145. doi: 10.1080/13623699.2021.1938035. Epub 2021 Jul 5. PMID 34225496

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial recruitment was done using referrals from key informants, community leaders, who were able to identify people affected by violence. To get more participants a snowball technique was used, participants were asked to refer others with similar problems. The identification numbers on the surveys were then randomized to one of the three arms.
Pre-assignment Details: 710 people were assessed for eligibility, 189 people were excluded: 175 for not meeting the inclusion criteria, 11 for meeting the exclusion criteria, and 3 refused to participate.
Groups:
- ARM 1: Common Elements Treatment Approach: Common Elements Treatment Approach (CETA) only
  Common Elements Treatment Approach: It was developed for treating symptoms related to violent trauma, i.e. symptoms of depression, anxiety and distress, among victimized population by violence and torture in Colombia. The most relevant components for treatment of these 3 problematic issues were identified from literature review and panel of experts. Descriptions and schemes have been developed in order to guarantee facility of use by community counselors who have little background in mental health skills. These counselors, who will be called Lay Psychosocial Community Workers (LPCW), will receive training in this technique before beginning of interventions. Application of this technique will be supervised constantly by mental health professionals (psychologist or social worker) from the project team.
- ARM 2: Narrative Community Group Therapy: Narrative Community Group Therapy (NCGT) only
  Community Therapy Intervention: It consists on teaching skills to people in the community to provide mental health therapy. Therapy will be performed by LPCW under constant supervision of mental health professionals (psychologists or social workers). Sessions will begin with a series of introductory activities that motivates participants to propose different problems that they would like to solve in the group. A participant proposed a problem and he/she will be asked to talk about it. LPCW and/or psychologist will support individuals if anyone needs help to solve a psychological crisis. At the end of this narration, participants will be asked about who has had a similar situation, and how they solved it. In this way, proposed solutions will be collected by the LPCW. Finally, session closes with a motivating activity.
- ARM 3: Standby Group: Standby group without intervention, but under monthly monitoring.
  Standby group: Standby group: they will be assessed at baseline with the initial survey and they will wait between 10 and 12 weeks; then an exit assessment will be performed with the study instrument. After the exit survey, control group participants will have an appointment with a professional psychologist to determine whether they require a mental health treatment. Those with such necessity will receive treatment in the ACOPLE center by professional psychologists or they will be referred to other health care level according to the type of psychopathology (e.g., psychosis) or its severity. Also, participants in the control group will be monitoring monthly by phone calls and if they have any psychological problem, they will be assessed in the ACOPLE center.
Period: Overall Study
Arm/Group | ARM 1: Common Elements Treatment Approach | ARM 2: Narrative Community Group Therapy | ARM 3: Standby Group
Started | 175 | 175 | 171
Buenaventura Participants | 92 | 89 | 88
Quibdó Participants | 83 | 86 | 83
Completed | 80 (A percentage of 75.1% completed the follow-up (exit survey)) | 90 (A percentage of 80.9% completed the follow-up (exit survey)) | 137
Not Completed | 95 | 85 | 34
Not completed — Withdrawal by Subject | 44 | 50 | 33
Not completed — Lost to Follow-up | 31 | 34 | 0
Not completed — Unknown reasons | 9 | 0 | 0
Not completed — Psychologist decision | 1 | 0 | 0
Not completed — Paperwork errors | 8 | 0 | 0
Not completed — Death | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ARM 1: Common Elements Treatment Approach: Common Elements Treatment Approach (CETA) only
  Common Elements Treatment Approach: It was developed for treating symptoms related to violent trauma, i.e. symptoms of depression, anxiety and distress, among victimized population by violence and torture in Colombia. The most relevant components for treatment of these 3 problematic issues were identified from literature review and panel of experts. Descriptions and schemes have been developed in order to guarantee facility of use by community counselors who have little background in mental health skills. These counselors, who will be called Mental Health Community Workers (MHCW), will receive training in this technique before beginning of interventions. Application of this technique will be supervised constantly by mental health professionals (psychologist or social worker) from the project team.
- ARM 2: Community Group Therapy: Community Group Therapy (CGT) only
  Community Therapy Intervention: It consists on teaching skills to people in the community to provide mental health therapy. Therapy will be performed by MHCW under constant supervision of mental health professionals (psychologists or social workers). Sessions will begin with a series of introductory activities that motivates participants to propose different problems that they would like to solve in the group. A participant proposed a problem and he/she will be asked to talk about it. MHCW and/or psychologist will support individuals if anyone needs help to solve a psychological crisis. At the end of this narration, participants will be asked about who has had a similar situation, and how they solved it. In this way, proposed solutions will be collected by the MHCW. Finally, session closes with a motivating activity.
- Total: Total of all reporting groups
Arm/Group | ARM 1: Common Elements Treatment Approach | ARM 2: Community Group Therapy | ARM 3: Standby Group | Total
Number analyzed (Participants) | 175 | 175 | 171 | 521
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 153 | 157 | 149 | 459
  >=65 years | 22 | 18 | 22 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Each row represents the studied population per city
  years
    Buenaventura: number analyzed (Participants) | 92 | 89 | 88 | 269
    Buenaventura | 40.4 (14.1) | 39.5 (13.3) | 41.8 (14.8) | 40.54 (14.08)
    Quibdó: number analyzed (Participants) | 83 | 86 | 83 | 252
    Quibdó | 46 (19) | 45.3 (29.5) | 44.3 (18.9) | 45.39 (19.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 157 | 150 | 456
  Male | 26 | 18 | 21 | 65
Region of Enrollment [Number; unit: participants]
  Colombia | 175 | 175 | 171 | 521

OUTCOME MEASURES:

1. Primary Outcome: Score Difference in Symptoms of Anxiety, Depression and Post-traumatic Stress Disorders.
Description: Symptoms, ranging from 0 for "never" to 3 for "all the time" being three the worst score, were assessed with adapted versions of Hopkins Symptom Checklist and Harvard Trauma Questionnaire. Constructs of depression (n=15 symptoms), anxiety (n=10 symptoms), and post-traumatic stress symptoms (n=16 symptoms) were extracted and analyzed out of the mentioned surveys. Depression and anxiety symptoms were assessed using the Hopkins Symptom Checklist (HSCL-25) and symptoms of trauma (PTSS) were assessed using the Harvard Trauma Questionnaire (HTQ).
  For each scale, the mean was calculated in order to use it as the measure for comparisons.
  Mean difference in scores of symptoms of anxiety, depression, and post-traumatic stress disorders between the subject's baseline and the final assessments were calculated.
Time Frame: Within the fifteen (15) days after finishing the intervention, either Common Elements Treatment Approach (CETA) or Narrative Community Group Therapy (NCGT). In the control group, 12 weeks after the baseline assessment.
Population: Each row represents participants per city
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- ARM 2: Narrative Community Group Therapy: Narrative Community Group Therapy (NCGT) only
  Narrative Community Therapy Intervention: It consists on teaching skills to people in the community to provide mental health therapy. Therapy will be performed by LPCW under constant supervision of mental health professionals (psychologists or social workers). Sessions will begin with a series of introductory activities that motivates participants to propose different problems that they would like to solve in the group. A participant proposed a problem and he/she will be asked to talk about it. LPCW and/or psychologist will support individuals if anyone needs help to solve a psychological crisis. At the end of this narration, participants will be asked about who has had a similar situation, and how they solved it. In this way, proposed solutions will be collected by the LPCW. Finally, session closes with a motivating activity.
Arm/Group | ARM 1: Common Elements Treatment Approach | ARM 2: Narrative Community Group Therapy | ARM 3: Standby Group
Number analyzed (Participants) | 175 | 175 | 171
units on a scale
  Buenaventura- Depression: number analyzed (Participants) | 92 | 89 | 88
  Buenaventura- Depression | -0.79 [-0.92 to -0.65] | -0.42 [-0.55 to -0.29] | -0.18 [-0.32 to -0.04]
  Quibdó- Depression: number analyzed (Participants) | 83 | 86 | 83
  Quibdó- Depression | -0.48 [-0.62 to -0.35] | -0.40 [-0.53 to -0.28] | -0.34 [-0.47 to -0.21]
  Buenaventura- Anxiety: number analyzed (Participants) | 92 | 89 | 88
  Buenaventura- Anxiety | -0.89 [-1.06 to -0.71] | -0.48 [-0.67 to -0.28] | -0.26 [-0.43 to -0.09]
  Quibdó- Anxiety: number analyzed (Participants) | 83 | 86 | 83
  Quibdó- Anxiety | -0.63 [-0.81 to -0.45] | -0.51 [-0.67 to -0.35] | -0.50 [-0.67 to -0.33]
  Buenaventura- Post Traumatic Stress: number analyzed (Participants) | 92 | 89 | 88
  Buenaventura- Post Traumatic Stress | -0.88 [-1.02 to -0.73] | -0.48 [-0.61 to -0.35] | -0.42 [-0.55 to -0.29]
  Quibdó- Post Traumatic Stress: number analyzed (Participants) | 83 | 86 | 83
  Quibdó- Post Traumatic Stress | -0.59 [-0.74 to -0.44] | -0.29 [-0.44 to -0.15] | -0.40 [-0.55 to -0.25]

2. Secondary Outcome: Score Difference in Total Mental Health Symptoms (TMHS) and Dysfunction
Description: TMHS scale of 64 items, ranging from 0 for "never" to 3 for "all the time" being the option three the worst condition, including locally relevant symptoms and sub-scales of depression (n=15 symptoms), anxiety (n=10 symptoms) and post-traumatic stress symptoms (PTSS) (n=16 symptoms). Depression and anxiety symptoms were assessed using the Hopkins Symptom Checklist (HSCL-25) and symptoms of trauma (PTSS) were assessed using the Harvard Trauma Questionnaire (HTQ).
  The Dysfunction measure was a gender-specific questionnaire with 12-items for females and 10-items for males. Each item assessed a task ranging from 0 for "no difficulty" to 4 for "cannot do it", being option four the worst condition.
  For each scale, the mean was calculated in order to use it as the measure for comparisons.
  Mean difference in scores of TMHS and Dysfunction between the subject's baseline and the final assessments were calculated.
Time Frame: as for outcome 1
Population: Each row represents participants per city
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ARM 1: Common Elements Treatment Approach | ARM 2: Narrative Community Group Therapy | ARM 3: Standby Group
Number analyzed (Participants) | 175 | 175 | 171
units on a scale
  Buenaventura- Total Mental Health Symptoms: number analyzed (Participants) | 92 | 89 | 88
  Buenaventura- Total Mental Health Symptoms | -0.74 [-0.85 to -0.63] | -0.39 [-0.50 to -0.29] | -0.28 [-0.38 to -0.18]
  Quibdó- Total Mental Health Symptoms: number analyzed (Participants) | 83 | 86 | 83
  Quibdó- Total Mental Health Symptoms | -0.49 [-0.60 to -0.39] | -0.35 [-0.46 to -0.23] | -0.38 [-0.49 to -0.26]
  Buenaventura- Dysfunction: number analyzed (Participants) | 92 | 89 | 88
  Buenaventura- Dysfunction | -0.41 [-0.56 to -0.26] | -0.31 [-0.50 to -0.14] | -0.01 [-0.18 to 0.15]
  Quibdó- Dysfunction: number analyzed (Participants) | 83 | 86 | 83
  Quibdó- Dysfunction | -0.08 [-0.26 to 0.1] | -0.29 [-0.46 to -0.11] | 0.002 [-0.18 to 0.18]

ADVERSE EVENTS:
Time Frame: The study time frame and 1 month after interventions follow-up
Description: Any untoward or unfavorable medical/psychological occurrence in a participant, including any abnormal sign, symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
  In every intervention session, follow-up calls (control group), and follow-up assessment, participants were asked about symptoms' changes, suicidal ideation, and other experienced issues.
Arm/Group | ARM 1: Common Elements Treatment Approach | ARM 2: Community Group Therapy | ARM 3: Standby Group
All-Cause Mortality (participants affected / at risk) | 1/175 | 1/175 | 0/171
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/175 | 0/171
Other Adverse Events (participants affected / at risk) | 0/175 | 0/175 | 0/171

LIMITATIONS AND CAVEATS:
This study will include a subsequent follow-up to assess middle-term effects of the interventions. The proportion of participants lost to follow-up represents a limitation. The low male participation in the study did not allow for a gender subgroup.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-10-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT01856673/Prot_SAP_000.pdf